CLINICAL TRIAL: NCT00302185
Title: A Feasibility Study in Acupuncture for Symptom Management in Palliative Care.
Brief Title: Acupuncture in Palliative Cancer Care
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Dr. Jan T. Lim, British Columbia Cancer Agency
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCCAVIC Pal 1
Record Dates: First submitted 2006-03-13; First posted 2006-03-14 (Estimated); Last update posted 2010-10-20 (Estimated); Status verified 2010-10

CONDITIONS: Neoplasms; Palliative Care
Keywords: Palliative Care; Acupuncture; Symptom Management; Quality of Life
MeSH Terms: conditions — Neoplasms | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nurse-led supportive care (Active Comparator): Visit with a Palliative Care nurse once weekly for 4 weeks
  Interventions: Behavioral: Nurse-led supportive care
- Acupuncture (Experimental): Patients received acupuncture once a week for 4 weeks.
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — Insertion of sterile, single-use acupuncture needles at 10-20 points including PC.6, HT.7, St.36, SP.6, and LR.3. Needles were connected to an electrical stimulator to mimick traditional manual stimulation with alternating patterns of stimulation for 20 minutes.
  Arms: Acupuncture
Behavioral: Nurse-led supportive care — 20-30 minutes of supportive attention from an experienced palliative nurse.
  Arms: Nurse-led supportive care

SUMMARY:
Research question: Can acupuncture improve symptom control and quality of life (QOL) in patients with advanced incurable cancer?

The purposes of this study is to investigate the feasibility of performing a randomized trial with acupuncture in improving symptom control and quality of life (QOL) in patients with advanced incurable cancer at the BC Cancer Agency, Vancouver Island Centre in Victoria.

We will:

* Evaluate whether subjects who are receiving palliative care for cancer related symptoms can tolerate and complete to a course of acupuncture treatments.
* Evaluate whether it is possible to conduct a study using acupuncture on cancer patients.

DETAILED DESCRIPTION:
Patients with advanced cancer suffer from many symptoms which dramatically reduce their Quality of Life (QOL). There have been significant improvements in the management of pain, nausea and constipation, but other common symptoms such as fatigue, anxiety, depression, and a lack of well-being are not readily addressed by conventional therapies. As cancer patients usually present with numerous symptoms, it would be important to try to address all of these globally, instead of only treating individual symptoms that respond well to conventional therapy. Attempts at controlling individual symptoms can also give rise to iatrogenic effects. One well known example is constipation occurring in patients who are on opiate analgesics. Successful treatment from the caregiver's perspective is often scored against each individual symptom that is being treated. From the patient's point of view, it is the interplay of the whole treatment package that succeeds or fails in improving his QOL

In an attempt at treating all of the patient's symptoms, research into the use of complementary and alternative medicine (CAM) has been conducted to determine the utility of these treatments in addressing the unmet needs of many patients with cancer. There is preliminary evidence that acupuncture in particular, is successful at improving many cancer and treatment associated symptoms.

Given the potential to improve symptom control and QOL, it is thought that acupuncture should be investigated to assess its effectiveness and feasibility in symptomatic patients with advanced cancer. Acupuncture should be compared against another intervention, so that the control group would also be receiving attention to their symptoms. As supportive care has been shown to be helpful in ameliorating symptoms in terminal care, acupuncture will be compared against this intervention. Sham acupuncture is not considered to be a good comparison for acupuncture as it is not well tested, and its effects are often indistinguishable from acupuncture. Recently however, some studies have reported the use of novel techniques that prevent acupuncture-naïve patients from distinguishing between acupuncture treatment and placebo. These techniques have yet to be independently validated.

Objectives: 1. To determine feasibility of recruiting patients and running a randomized study that involves acupuncture at the BCCA-VIC. 2. To gather enough data to support a grant application to fund a larger study to look at the effectiveness of acupuncture as adjunctive treatment for the management of symptoms associated with palliative cancer care.

ELIGIBILITY:
Inclusion Criteria:

* patients receiving palliative therapy for incurable cancer
* anticipated survival of at least 3 months
* able to complete ESAS sheet unaided
* ESAS of 5 or more in at least one of the following symptoms; fatigue, depression, anxiety and lack of wellbeing

Exclusion Criteria:

* refuse to receive weekly acupuncture for 4 weeks
* refuse to receive nursing support for 4 weeks
* known to have impaired clotting of blood

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-06; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
The change in Edmonton Symptom Assessment Score (ESAS) after intervention (ESAS at baseline - ESAS at first follow up) will be analysed for each of the 4 symptoms (fatigue, anxiety, depression, a lack of well-being) under investigation. Results will be

SECONDARY OUTCOMES:
Determine the % of patients suitable, and the % of patients who consent to be recruited.
Determine the % of patients who complete all 4 intervention sessions.
Determine the duration of change in ESAS after intervention (ESAS at second and third follow-up - ESAS at first follow up).

CONTACTS AND LOCATIONS:
Overall Officials: Jan T Lim, MD, Principal Investigator — BC Cancer Agency and University of British Columbia
Locations (1):
- BC Cancer Agency - Vancouver Island Centre, Victoria, British Columbia, Canada